CLINICAL TRIAL: NCT07278661
Title: Preoperative Use of Romiplostim in Thrombocytopenic Patients Undergoing Cardiac Surgery. A Phase 3, Multicenter Randomized Double-blinded Controlled Against Placebo Study.
Brief Title: Preoperative Use of Romiplostim in Thrombocytopenic Patients Undergoing Cardiac Surgery.
Acronym: CT-PLATE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC24_0458; 2024-517710-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chirurgical Intervention; Thrombocytopaenia
Keywords: Thrombocytopenia; Cardiac Surgery; Growth Factor; Patient Blood Management
MeSH Terms: conditions — Thrombocytopenia | interventions — romiplostim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Romiplostim (Experimental): injection sc
  Interventions: Drug: Nplate
- NaCl (Placebo Comparator): injection sc
  Interventions: Drug: NaCl %0.9

INTERVENTIONS:
Drug: Nplate — The dosage for this first injection will be:
  * 2 µg/kg for patients with a platelet count at inclusion between 149,000 and 100,000/mm3
  * 3 µg/kg for patients with a platelet count strictly below 100,000/mm3
  Arms: Romiplostim
Drug: NaCl %0.9 — NaCl (Sodium chloride) 0.9% administered subcutaneously
  Arms: NaCl

SUMMARY:
Romiplostim has demonstrated its efficacy and good tolerance in multiple indications. If the efficacy of Romiplostim is confirmed in this population, thrombocytopenic patients will be able to undergo cardiac surgery, which is generally life-saving, without prior thrombocytopenia.

Patients included in the study will be hospitalized within 15 days of the first administration of the study treatment and will be closely monitored clinically and biologically for at least 10 days after surgery. The occurrence of an adverse event can therefore be quickly detected and managed.

Collectively, "Patient Blood Management" strategies are mainly focused on the management of preoperative anemia. If positive, this study will enrich the therapeutic arsenal available for optimizing patients in preparation for major surgery. As no major collective complications are expected, the collective benefit/risk ratio also appears favorable.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with no upper age limit,
* Scheduled cardiac surgery with cardiopulmonary bypass,
* Patients with preoperative thrombocytopenia strictly <150,000/mm3
* Surgery performed with a blood recovery system using centrifugation (Cell Saver type) or equivalent,
* Feasibility of a first injection (Romiplostim or Placebo) between D-14 and D-10 before surgery,
* Surgery requiring the administration of antiplatelet and/or anticoagulant therapy for a minimum of 1 month postoperatively.

Exclusion Criteria:

* Inability to administer the first injection of Romiplostim or Placebo within 10 days prior to surgery,
* Cardiac surgery without cardiopulmonary bypass,
* Coronary artery bypass grafting due to one or more significant coronary stenoses,
* Tangential filtration blood recovery system (i-SEP SAME® type) planned for intraoperative use or absence of intraoperative blood recovery system due to investigator choice or availability issues,
* Planned use of aprotinin as an antifibrinolytic agent during surgery,
* Patient with contraindication to discontinuation of all antiplatelet therapy before surgery (with discontinuation at least 3 days before surgery for acetylsalicylic acid and at least 5 days before surgery for clopidogrel/ticagrelor),
* Hereditary or acquired thrombophilia with or without a history of thrombosis,
* History of ischemic or hemorrhagic stroke,
* History of phlebitis, pulmonary embolism, or portal vein thrombosis,
* History of heart attack with stent placement less than one year ago,
* Current limb immobilization (e.g., plaster cast for ankle fracture) or inability to walk independently due to limited mobility (e.g., paralysis),
* Current immobilization of a limb (e.g., plaster cast for ankle fracture) or inability to walk independently due to motor limitation (e.g., complete paralysis of a limb) or medical contraindication (e.g., strict bed rest required),
* Myelogram indicating malignant hematological disease or blast cells strictly greater than 5%,
* Malignant diseases with last follow-up indicating disease progression,
* Severe chronic liver disease with a CHILD-PUGH score > 6 (measured without decompensation),
* Treatment with thrombopoietin receptor agonist received within 3 months prior to inclusion,
* Treatment with JAK2 inhibitor currently underway or within the last month,
* Treatment with Rituximab within the last 7.5 months or intravenous immunoglobulin within the last 40 days,
* Ongoing treatment with corticosteroids at doses equal to or greater than 20mg of hydrocortisone, 5mg of prednisone/or prednisolone, 4mg of methylprednisone, or 0.75mg of dexamethasone,
* Known hemophilia,
* Hypersensitivity to romiplostim or any of its excipients, or to proteins derived from E. coli,
* Context of hyperchloremia, hypernatremia, or major water and salt retention with anasarca refractory to medical treatment,
* Pregnant women or women of childbearing age who are not using effective contraception,
* Currently using combined oral contraceptive pills or oral hormone replacement therapy containing estrogen,
* Breastfeeding women,
* Minors,
* Adults under guardianship, curatorship, or judicial protection,
* Patients who do not speak French,
* Patients without Social Security coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Day 7
  Lowest platelet count measured between the end of ECC and the 7th postoperative day with D0 = day of surgery

SECONDARY OUTCOMES:
Transfusion of platelet concentrate | Day 1
  Number of transfusion of platelet concentrate
Transfusion of platelet concentrate | Day 7
  Number of transfusion of platelet concentrate
Transfusion of platelet concentrate | Day 28
  Number of transfusion of platelet concentrate
Transfusion of red blood cell concentrate | Day 1
  Number of transfusion of red blood cell concentrate
Transfusion of red blood cell concentrate | Day 7
  Number of transfusion of red blood cell concentrate
Transfusion of red blood cell concentrate | Day 28
  Number of transfusion of red blood cell concentrate
Transfusion of fresh frozen plasma | Day 1
  Number of transfusion of fresh frozen plasma
Transfusion of fresh frozen plasma | Day 7
  Number of transfusion of fresh frozen plasma
Administration of blood-derived drugs | Day 1
  Number of administration of blood-derived drugs
Administration of blood-derived drugs | Day 7
  Number of administration of blood-derived drugs
Administration of blood-derived drugs | Day 28
  Number of administration of blood-derived drugs
Efficacy | Day 28
  Lowest platelet count measured between the end of ECC and the 28th postoperative day with D0 = day of surgery
Efficacy | Day 7
  Highest platelet count measured between the end of ECC and the 7th postoperative day with D0 = day of surgery
Efficacy | Day 28
  Highest platelet count measured between the end of ECC and the 28th postoperative day with D0 = day of surgery
Lowest haemoglobin | Day 7
  Lowest haemoglobincount measured between the end of ECC and the 7th postoperative day with D0 = day of surgery
Lowest haemoglobin | Day 28
  Lowest haemoglobincount measured between the end of ECC and the 28th postoperative day with D0 = day of surgery
Bleeding volume | Hour 12
  Post-operative bleeding volume from sternal closure to 12th post-operative hour
Bleeding volume | Day 1
  Post-operative bleeding volume from sternal closure to 24th post-operative hour
Mortality | Day 28
  Rate of mortality
Infection | Month 3
  Rate of infection

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Dijon, Dijon
  - CHU de Nantes, Nantes
  - Hôpital Bichat (AP-HP), Paris
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg